CLINICAL TRIAL: NCT05791487
Title: Remission With Diet for Ulcerative Colitis Exacerbations: A Single Blinded, International Randomized Controlled Clinical and Translational Trial
Brief Title: Combination of Diet and Oral Budesonide for Ulcerative Colitis
Acronym: ReDUCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0073-22-WOMC
Record Dates: First submitted 2023-02-16; First posted 2023-03-30 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Chronic Mild; Ulcerative Colitis Chronic Moderate
Keywords: Ulcerative colitis; Diet; Partial enteral nutrition; Microbiome
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Budesonide

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulcerative colitis Exclusion Diet + Partial enteral nutrition (Experimental): Participants in Group 1 will receive the UCED combined with partial enteral nutrition (PEN) using a novel nutritional formula for 6 weeks (diet phase 1) that will add to oral budesonide 9 mg topical therapy for 6 weeks and will follow diet + PEN (phase 2: wk6-wk12) and diet phase 3 for 24 weeks.
  Interventions: Other: Ulcerative colitis Exclusion Diet; Other: Partial enteral nutrition (PEN); Drug: Oral Budesonide
- Free diet (Active Comparator): Participants in Group 2 will receive oral budesonide 9 mg topical therapy alone for 6 weeks with no dietary intervention
  Interventions: Other: free diet; Drug: Oral Budesonide

INTERVENTIONS:
Other: Ulcerative colitis Exclusion Diet — a limited whole food diet (UCED)
  Other Names: UCED
  Arms: Ulcerative colitis Exclusion Diet + Partial enteral nutrition
Other: Partial enteral nutrition (PEN) — The diet will be supplemented by 3 glasses a day (750 m"l) of the formula developed for UC using the UCED principles.
  Other Names: UC nutritional formula, Nestle
  Arms: Ulcerative colitis Exclusion Diet + Partial enteral nutrition
Other: free diet — oral Budeosnide for 6 weeks + free diet
  Arms: Free diet
Drug: Oral Budesonide — Oral Budesonide 9 mg

SUMMARY:
The ReDUCE Trial is a multinational single-blinded randomized controlled trial in mild to moderate flare of Ulcerative colitis (UC) disease patients. The purpose of the study is to validate the clinical efficacy of the UCED (Ulcerative colitis Exclusion Diet) with partial enteral nutrition (PEN) using a novel formula.

The investigators anticipate that adding a novel specifically designed dietary intervention in addition to drug will lead to superior remission and mucosal healing via changes in the microbiome.

DETAILED DESCRIPTION:
Rational: Ulcerative colitis is currently treated only by medical therapies or surgery and there is no other option to avoid immune suppression.

Thus, developing a dietary therapy that would treat the cause of the disease, while having no side effects, would likely lead to immediate implementation and be sought out by patients hesitant to be on lifelong medications or immune suppression.

Objectives: To evaluate if the UC Exclusion Diet (UCED), can improve outcomes when administered with an oral budesonide regimen to adult patients with mild to moderate UC.

Methods: This will be a 24-week multinational single-blinded randomized controlled trial.

After a baseline flexible sigmoidoscopy, Group 1 will receive oral budesonide 9 mg topical therapy + the UCED+PEN phase 1 diet for 6 weeks, while Group 2 will receive oral budesonide 9 mg topical therapy alone for 6 weeks with no dietary intervention.

Both groups will continue the previous maintenance therapy through week 12 and both groups will stop budesonide at week 6.

Group 1 will continue with the phase 2 diet/PEN from week 7-12 while group 2 will stay on habitual diet. A flexible sigmoidoscopy will be repeated at week 12.

Population: adults and adolescents between the ages of 17-65 with a mild to moderate active disease (Simple Clinical Colitis Activity Index (SCCAI) 5-10 with an endoscopic Mayo score 1-3), on an existing maintenance therapy comparing two arms.

Time frame: The induction of remission phase will last 8 weeks followed by maintenance phase for a period of 24 weeks

Expected outcomes and significance: The investigators anticipate that adding a novel specifically designed dietary intervention in addition to drug will lead to superior remission and mucosal healing via changes in the microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Established diagnosis of UC with mild to moderate active disease, 5 ≤ SCCAI ≤ 10
* Age: 17-65 years (inclusive)
* Extent E1-E3 by the Montreal classification
* Active colitis in the rectum or sigmoid colon on sigmoidoscopy
* Stable medication use of oral 5ASA for at least 8 weeks, thiopurines, vedolizumabs, Ustekinumab or tofacitinib for at least 12 weeks

Exclusion Criteria:

* Severe colitis (SCCAI>10) hospitalization for acute severe colitis (ASC) in the previous 6 months
* Use of steroids in the previous 3 months
* Patients treated with Anti-TNF currently or in patients who had previously failed or lost response to anti TNF
* Vegans (vegetarians may enroll)
* Pregnancy
* Inability use of budesonide due to severe adverse events
* Extraintestinal manifestations such as arthritis, spondyloarthropathy or uveitis
* Presence of baseline hypoalbuminemia
* Fever >38°C
* Evidence for Clostridioides difficile infection
* Renal failure
* Hepatitis or PSC (Primary Sclerosing Cholangitis)
* Active malignancy (excluding skin BCC).

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Steroid free remission | week 12
  Steroid free intention-to-treat (ITT) remission according to SCCAI<3 at week 12
  *The Simple Clinical Colitis Activity Index (SCCAI). score ranges from 0 to 19. clinical remission will be defined according to SCCAI<3

SECONDARY OUTCOMES:
Clinical response | week 12
  *The Simple Clinical Colitis Activity Index (SCCAI). score ranges from 0 to 19 . Clinical response defined as 3-point reduction in SCCAI or remission.
Steroids free remission | week 6
  Steroid free intention-to-treat (ITT) remission according to SCCAI<3 at week 6
  *The Simple Clinical Colitis Activity Index (SCCAI). score ranges from 0 to 19. clinical remission will be defined according to SCCAI<3
Sustained steroid free remission | week 24
  according to SCCAI<3 at week 24 score ranges from 0 to 19. clinical remission will be defined according to SCCAI<3
Endoscopic remission | week 12
  Defined as Mayo score 0 or 1. Mayo score 0 or 1 means endoscopic remission.
  *The Mayo Score for ulcerative colitis disease activity provides an assessement of disease severity and can be used to monitor patients during therapy.
Change in medical therapy | by week 12
  Need for additional or change in medical therapy according to the physician decision.
Fecal calprotectin | week 12
  Fecal calprotectin will be analyzed locally, and will be defined as median/mean change in calprotectin from baseline.

CONTACTS AND LOCATIONS:
Locations (6):
- Israel (3):
  - Emek Medical Center, Afula
  - Wolfson Medical Center, Holon
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- FONDAZIONE GEMELLI HOSPITAL Catholic University of the Sacred Hearth, Roma, Italy
- Radboud University Medical Center (Radboudumc), Nijmegen, Netherlands
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarbagili Shabat C, Scaldaferri F, Zittan E, Hirsch A, Mentella MC, Musca T, Cohen NA, Ron Y, Fliss Isakov N, Pfeffer J, Yaakov M, Fanali C, Turchini L, Masucci L, Quaranta G, Kolonimos N, Godneva A, Weinberger A, Kopylov U, Levine A, Maharshak N. Use of Faecal Transplantation with a Novel Diet for Mild to Moderate Active Ulcerative Colitis: The CRAFT UC Randomised Controlled Trial. J Crohns Colitis. 2022 Mar 14;16(3):369-378. doi: 10.1093/ecco-jcc/jjab165. PMID 34514495
- [Background] Sarbagili-Shabat C, Albenberg L, Van Limbergen J, Pressman N, Otley A, Yaakov M, Wine E, Weiner D, Levine A. A Novel UC Exclusion Diet and Antibiotics for Treatment of Mild to Moderate Pediatric Ulcerative Colitis: A Prospective Open-Label Pilot Study. Nutrients. 2021 Oct 23;13(11):3736. doi: 10.3390/nu13113736. PMID 34835992
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34514495/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34835992/